CLINICAL TRIAL: NCT01007513
Title: Cervical Assessment by Supracervical, Cervical and Vaginal Markers: Simultaneous Transvaginal Ultrasound and Inflammatory Proteins Detection
Brief Title: Study of Cervix and Inflammation in Preterm Birth Prediction
Acronym: COLIBRI
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-Charles Pasquier, Dr, Université de Sherbrooke
Other Study IDs: 08-020
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Preterm Birth
Keywords: Prematurity; Inflammation; Transvaginal ultrasound; Vaginal secretion; Inflammatory process; Neonatal morbidity
MeSH Terms: conditions — Premature Birth; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal secretion
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- At risk patient for preterm delivery: Patient referred to the MFM clinic for a risk evaluation for preterm delivery.
  Interventions: Procedure: Transvaginal ultrasound; Procedure: Vaginal secretion sampling

INTERVENTIONS:
Procedure: Transvaginal ultrasound — A transvaginal ultrasound with an endocavitary probe will be done as required by the medical condition of the patient. The cervical and supracervical factors will be noted.
Procedure: Vaginal secretion sampling — Vaginal secretion swab will be collected each time patient will have a transvaginal ultrasound. The sample will be centrifuged, frozen and store to be analysed at the end of the study with multiplex antibody arrays.
  Other Names: Ray Biotech Multiplex Antibody Arrays

SUMMARY:
Preterm birth rate is 7.2% in Quebec, it's risen worldwide in the past decade and it's the leading cause of perinatal mortality and morbidity. Preterm birth is a major public health problem. Preterm labor leading to preterm birth is difficult to diagnose and prediction of preterm birth is a medical challenge. In the past years, research found that transvaginal ultrasound to assess the cervix of the uterus and vaginal detection of inflammatory protein, specific bacteria and fetal fibronectin can help to detect women at increase risk of preterm delivery. The investigators believe that a combination of these tests can lead to a better prediction of preterm delivery. The investigators want to conduct a study among women judged at increase risk of preterm delivery by their physician (having contractions, modified cervix, past-history of preterm delivery or multiple pregnancy) and assess their cervix by ultrasound and sample their vaginal secretion. The investigators want to analyze the vaginal sampling and look for inflammatory proteins. The objective of this study is to prove the feasibility of this assessment method and elaborate a better predictive test that the investigators can easily use in obstetrics clinics and hospitals.

DETAILED DESCRIPTION:
Preterm birth rate in Quebec is 7.2% and, despite extensive research, the rate of preterm birth has risen worldwide over the past decades. Preterm birth is, all over the world, the first cause of perinatal mortality and morbidity. Spontaneous preterm birth (sPTB) groups premature births with intact and ruptured membranes and represents 70% of preterm delivery. The two conditions associated with sPTB share a common physiopathology and a progressive cascade of events. Extensive evidence supports a central role for the production of prostaglandins, inflammatory cytokines and matrix metalloproteinases (MMP) in the cervix and decidua to promote cervical ripening and decidual and fetal membrane activation but, the exact progression of events remains unclear. Several factors were described as risk factor for sPTB like bacterial vaginosis, inflammatory cytokines and fetal fibronectin in vaginal secretions. The transvaginal ultrasound of the cervix (TVUS), which estimates the length and the aspect of the cervix, can be used as predictive factor of preterm birth. To date, no study has addressed the supra-cervical region by transvaginal ultrasound. This region may be an important key of the inflammatory process leading to sPTB. The assessment of this region by ultrasound can be a predictive marker of sPTB. We want to prove the feasibility of this new approach of sPTB prediction : the transvaginal ultrasound assessment of the supracervical and cervical region associated with detection of vaginal inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Live singleton or multiple pregnancy
* Clinical risk of preterm delivery
* Pregnancy between 20 and 34 gestational weeks

Exclusion Criteria:

* Delivery on the day of the ultrasound
* Major fetal anomaly
* Previa placentation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: At risk women referred by their physician to the MFM clinic for evaluation of preterm birth risk.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Preterm birth < 34 gestational weeks among patient with presence of supracervical factor at ultrasound study. | December 2009

SECONDARY OUTCOMES:
Presence of inflammatory proteins in vaginal secretion of patient with presence of supracervical factors at transvaginal ultrasound. | December 2009
Neonatal morbidity of preterm infant. | December 2009

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, Md, PhD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Raiche E, Ouellet A, Berthiaume M, Rousseau E, Pasquier JC. Short and inflamed cervix predicts spontaneous preterm birth (COLIBRI study). J Matern Fetal Neonatal Med. 2014 Jul;27(10):1015-9. doi: 10.3109/14767058.2013.847917. Epub 2013 Nov 14. PMID 24228627